CLINICAL TRIAL: NCT06676241
Title: One-stage and Delayed Laparoscopic Cholecystectomy After Endoscopic Retrograde Cholangiopancreatography with Endoscopic Sphincterotomy in Cholecystocholedocholithiasis
Status: Completed | Type: Observational
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16/17.10.2024
Record Dates: First submitted 2024-10-27; First posted 2024-11-06 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Choledocholithiasis; Cholecystolithiasis; Cholangiopancreatography, Endoscopic Retrograde; Laparoscopic Cholecystectomy; Children; Acute Pancreatitis (AP); Common Bile Duct Calculi
Keywords: Сholedocholelysis; Endoscopic retrograde cholangiopancreatography (ERCP)
MeSH Terms: conditions — Choledocholithiasis; Cholecystolithiasis; Pancreatitis; Gallstones | interventions — Cholangiopancreatography, Endoscopic Retrograde; Cholecystectomy, Laparoscopic; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ERCP, EST and simultaneous LC: Patients aged 10-80 years initially underwent ERCP with ES by an endoscopist with the consent of the patient or legal representative. Patients underwent endoscopic procedures using fluoroscopy in the operating room, under general anesthesia. Laparoscopic cholecystectomy was performed immediately after ERCP with ES under general anesthesia
  Interventions: Procedure: endoscopic retrograde cholangiopancreatography; laparoscopic cholecystectomy
- ERCP, EST and LC in a delayed manner: Patients aged 0-17 years initially underwent ERCP with ES by an endoscopist with the consent of the patient or legal representative. Patients underwent endoscopic procedures using fluoroscopy in the operating room, under general anesthesia. Laparoscopic cholecystectomy was performed in a delayed manner, not earlier than 7 days after ERCP
  Interventions: Procedure: endoscopic retrograde cholangiopancreatography;laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: endoscopic retrograde cholangiopancreatography; laparoscopic cholecystectomy — Initially, ERCP with EST was performed by an endoscopist with the consent of the patient or legal representative. The patients underwent endoscopic procedures using fluoroscopy in the operating room, under general anesthesia. Subsequently, laparoscopic cholecystectomy was performed immediately after ERCP with ES under general anesthesia.
  Other Names: Cholangiopancreatography; Laparoscopic
  Groups: ERCP, EST and simultaneous LC
Procedure: endoscopic retrograde cholangiopancreatography;laparoscopic cholecystectomy — Initially, ERCP with EST was performed by an endoscopist with the consent of the patient or legal representative. The patient underwent the endoscopic procedure using fluoroscopy in the operating room, under general anesthesia. Subsequently, laparoscopic cholecystectomy was performed on a delayed basis no earlier than 7 days after ERCP
  Other Names: Cholangiopancreatography; Laparoscopic
  Groups: ERCP, EST and LC in a delayed manner

SUMMARY:
In this study, it is planned to compare ERCP with ES + delayed LC in children, with one-stage LC + ERCP with ES in adults to confirm that ERCP with ES + delayed LC is more suitable for pediatric patients with cholecystocholedocholithiasis.

DETAILED DESCRIPTION:
Nowadays there is no gold standard for the treatment of choledocholithiasis combined with cholecystolithiasis in the pediatric population. The most common method for resolving the biliary obstruction is endoscopic retrograde cholangiopancreatography (ERCP) with endoscopic sphincterotomy (EST) and laparoscopic cholecystectomy (LC). In the adult practice, the approaches to the treatment of choledocholithiasis include the following items: laparoscopic common bile duct exploration (LCBDE), laparoendoscopic rendezvous method (LERV) and LC after ERCP. Both LCBDE and LERV allow for the simultaneous treatment of cholecystocholedocholithiasis. However, a great number of medical institutions do not have an opportunity to use these methods due to the difficulties of implementation and the need for special training and experience of specialists. The timing of LC after ERCP in patients with cholecystocholedocholithiasis also remains a subject of debate. Numerous studies recommend early LC after ERCP. However, there are high risks of injury to the common bile duct and hepatic vessels against the background of acute inflammatory process in the area of hepatoduodenal ligament. In this study, it is planned to compare ERCP with ES + delayed LC in children, with one-stage LC + ERCP with ES in adults to confirm that ERCP with ES + delayed LC is more suitable for pediatric patients with cholecystocholedocholithiasis.

The aim of this study is to evaluate the efficacy and safety of endoscopic retrograde cholangiopancreatography, endoscopic sphincterotomy with delayed laparoscopic cholecystectomy in children with cholecystocholedocholithiasis compared with one-stage cholangiopancreatography, endoscopic sphincterotomy and laparoscopic cholecystectomy in adults with cholecystocholedocholithiasis.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from the patient, child or legal representative
* Age 0-80 years
* Acute cholecystitis
* Choledocholithiasis
* Intraoperative ERCP
* Preoperative ERCP followed by cholecystectomy

Exclusion Criteria:

* Unwillingness or inability to consent to the study
* Pregnancy
* Age > 80 years
* Previous ERCP or percutaneous transhepatic biliary drainage
* Anastomosis in the upper gastrointestinal tract
* Benign or malignant stricture
* Preoperative comorbidities: gastrointestinal bleeding, severe liver disease, acute and chronic cholangitis, other known cholestatic hepatopancreatobiliary disease, septic shock.
* In combination with Mirizzi syndrome and intrahepatic bile duct stones
* Congenital anomaly of the biliary tract
* Malignant neoplasms
* Acute pancreatitis

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Recurrence of stones in the common bile duct | 30 days after ERCP
  The diagnosis of the stone in the common bile duct.

SECONDARY OUTCOMES:
Bleeding | 30 days after ERCP
  decreased hemoglobin level, visual picture during endoscopic examination, positive stool for occult blood
Perforation | 30 days after ERCP
  by CT, radiography (fluid or gas in the retroperitoneal space or abdominal cavity, visual picture during endoscopic examination)
Bile leak | 30 days after ERCP
  bile aspirated from the abdominal cavity
Acute cholangitis | 60 days after ERCP
  intermittent chills, fever, increased proinflammatory blood markers after ERCP
Bile duct stricture | 1 year after ERCP
  after ERCP
Time spent in hospital until discharge | from admission to hospital until the end of treatment (up to 8 weeks)
Technical success - success of the procedures as documented by a yes or no | 1 month
Duration of the laparoscopic cholecystectomy,min | From enrollment to the end of treatment (3 month)
Acute pancreatitis | within 14 days after ERCP
  at least two out of three criteria according to the classification developed by the INSPPIRE group
Duration of the Endoscopic retrograde cholangiopancreatography | From enrollment to the end of treatment (3 month)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy А Pyhteev, PhD, Study Director — Head of the Department of Pediatric Surgery; Leonid M Elin, Principal Investigator — Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky
Locations (1):
- Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky, Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
A complete dataset can be provided upon reasoned request